CLINICAL TRIAL: NCT06563765
Title: FAP-targeting PET/CT for Noninvasive Monitoring of Renal Fibrosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-386
Record Dates: First submitted 2024-06-02; First posted 2024-08-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-07

CONDITIONS: CKD; Renal Fibrosis
Keywords: CKD; Renal fibrosis; FAP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAP-targeting PET/CT imaging (Experimental): FAP-targeting PET/CT imaging will be performed on the enrolled patients.
  Interventions: Other: FAP-targeting PET/CT imaging will be performed on the enrolled patients.

INTERVENTIONS:
Other: FAP-targeting PET/CT imaging will be performed on the enrolled patients. — FAP-targeting PET/CT imaging will be performed on the enrolled patients.

SUMMARY:
Chronic kidney disease (CKD) is an irreversible change of kidney function and structure caused by many reasons. The main threat of CKD to human health is progressive renal function decline. Delaying the progression of chronic kidney disease to end-stage renal failure is an important clinical need, and renal fibrosis is a common pathway for the progression of chronic kidney disease to end-stage renal failure. The evaluation of renal fibrosis is of great value for the course and prognosis of patients with chronic kidney disease. However, pathological detection has the disadvantages of trauma, false negative, and cannot be implemented repeatedly. At present, there is a lack of effective non-invasive, dynamic, real-time monitoring and evaluation means. A commercially available FAP-targeted imaging agent, FAPI-04, has been used for PET/CT imaging of systemic fibrosis lesions with high uptake background in normal kidneys. Although it can show severe renal fibrosis, it is not conducive to the detection rate of patients with mild-moderate fibrosis who need more accurate evaluation. The new targeted FAP imaging agent successfully constructed by our research group has proved that it can show the degree of renal fibrosis at the living level and has correlation. Therefore, this study intends to carry out a series of clinical studies on the imaging of renal fibrosis with new targeted FAP probes, evaluate the specificity and sensitivity of the new targeted FAP probes in the diagnosis of renal fibrosis, and ultimately provide a new method for clinical dynamic, non-invasive assessment and monitoring of the degree and progression of renal fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease
* Renal pathology was performed within 2 weeks

Exclusion Criteria:

* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Pathological type | 1 week after enrollment
  pathological type (e.g., sclerosing IgA nephropathy)
Baseline serum creatinine (μmol/L) | 1 month before enrollment and 1 month after enrollment
  laboratory results
Baseline 24-hour urinary protein (g/24h) | 1 month before enrollment and 1 month after enrollment
  laboratory results
Quantified renal pathological involvement. | 1 week after enrollment
  Based on kidney biopsy sections, interstitial atrophy, interstitial inflammatory infiltration, and tubular fibrosis will be quantified.
Pathological MESTC score | 1 week after enrollment
  MESTC score (0-2, for IgA nephropathy patients)

SECONDARY OUTCOMES:
Follow-up serum creatinine (μmol/L) | From 1 month after enrollment to 60 month after enrollment
  laboratory results
Proteinuria remisssion | From 1 month after enrollment to 60 month after enrollment
  For IgA nephropathy (IgAN) patients with baseline urinary total protein (UTP) exceeding 0.5 g/24h, a reduction of UTP to below 0.5 g/24h without recurrence within 4 weeks was considered proteinuria remission.
Acute kidney disease remission | Within 3 month after enrollment
  For IgAN patients with AKD, AKD remission was defined as a reduction in SCr to below 75% of the peak value within 90 days after imaging. Remission was classified as complete if the difference between the last recorded SCr and baseline SCr was ≤26.5 μmol/L; otherwise, it was classified as partial. Baseline SCr was defined as the lowest value recorded within 90 days prior to hospital admission. If unavailable, the lowest SCr value within 90 days after admission was used as the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China